CLINICAL TRIAL: NCT02125500
Title: Pilot Study to Assess Efficacy and Safety of Sofosbuvir/Ledipasvir (GS-5885) Fixed-dose Combination in NS3/4A Protease Inhibitor-experienced Subjects With HCV Genotype 1 Infection and HIV Co-infection
Brief Title: Pilot Study to Assess Efficacy and Safety of Sofosbuvir/Ledipasvir Fixed-dose Combination in Treatment Experienced Subjects With Hepatitis C Virus (HCV) Genotype 1 - HIV Co-infection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ANRS HC31 SOFTRIH
Record Dates: First submitted 2014-04-24; First posted 2014-04-29 (Estimated); Last update posted 2017-06-29 (Actual); Status verified 2017-06

CONDITIONS: Viral Hepatitis C; HIV
Keywords: HCV/HIV coinfection; HCV genotype 1
MeSH Terms: conditions — Hepatitis C | interventions — Sofosbuvir; ledipasvir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Sofosbuvir/Ledipasvir (Experimental): Non-cirrhotic patients will receive SOF/LDV Fixed Dose Combination (FDC) for 12 weeks.
  Cirrhotic patients will receive SOF/LDV Fixed Dose Combination (FDC) for 24 weeks.
  Interventions: Drug: Sofosbuvir/Ledipasvir fixed dose

INTERVENTIONS:
Drug: Sofosbuvir/Ledipasvir fixed dose — SOF 400 mg/LDV 90 mg FDC tablet administered orally once daily
  Other Names: Sofosbuvir is also known as GS-7977 or PSI-7977.; Ledipasvir is also known as GS-5885.

SUMMARY:
Aim of the study is to assess the efficacy and safety of 24 weeks of oral Sofosbuvir/Ledipasvir fixed-dose combination (FDC) in subjects with HCV genotype 1 infection and HIV co-infection, who have previously failed a NS3/4A protease inhibitor plus Pegylated interferon /ribavirin regimen or stopped prematurely their treatment for intolerance.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed HIV infection
* Infection with HCV genotype 1 only, confirmed at screen visit, with a HCV-RNA ≥ 1000 InternationalUnit(IU)/mL at screen visit
* Treatment-experienced subjects with:
* previous virological failure to tritherapy with Peginterferon/Ribavirin and protease inhibitor,
* or premature discontinuation of previous tritherapy with Peginterferon/Ribavirin and protease inhibitor due to intolerance to Peginterferon or protease inhibitor
* Anti-HCV treatment stopped for at least the last 3 months
* Patients on a stable (for more than 1 month) antiretroviral treatment consisting of an emtricitabine/tenofovir or lamivudine/tenofovir standard of care backbone plus efavirenz or raltegravir or rilpivirine or enfuvirtide. Alternative combinations of the above listed medications may be allowed.
* Dendritic cells 4 > 100/mm3 and > 15% at screen visit
* HIV-RNA < 50cp/ml for more than 3 months at screen visit
* Any liver fibrosis grade, with the assessment of the presence or not of cirrhosis at screening, cirrhosis being defined as a METAVIR score of F4 on the liver puncture biopsy and/or with hepatic impulse elastometry ≥ 14,5 kilopascal (kPa):
* Previous liver biopsy exhibiting cirrhosis lesions (METAVIR F4),

  * and/or significant liver biopsy (cumulative length ≥ 15mm or ≥ 5 portal spaces), within the past 18 months
  * and/or significant and reliable liver stiffness assessment (Fibroscan®) within the past 6 months (at least 10 measures with IQR less than 30% of the median value and a success rate of at least 70%).
* Female patients with child-bearing potential, and their heterosexual partners must use adequate contraception from the date of screening until 90 days after administration of the last dose of study drug. Male participants must agree to consistently and correctly use a condom, while their female partner must use adequate contraception from the date of screening until 90 days after administration of the last dose of study drug
* Body weight ≥40 kg and ≤125 kg
* Informed and signed consent for the main study and the Pharmacokinetic (PK ) sub-study (for the participating patients)
* Patients with Health insurance

Non inclusion Criteria:

* Child-Pugh B or C cirrhosis or history of decompensated cirrhosis.
* Co-infection with Hepatitis B virus (HBV) (AgHBs +) with HBV DNA > 1000 UI/ml
* Pregnant or breast-feeding women
* Transplant recipients
* Opportunistic infections (stage C), active or occurred within 6 months prior to baseline
* Evolutive malignancy, including hepatocarcinoma which should be controlled prior to baseline
* Alcohol or drug consumption which may affect the study participation according to the investigator. Patients included in a programme of substitution with methadone or buprenorphine could be enrolled. The opinion of a consultant in addictology is recommended for patients presenting with current drug use or drug use during the previous year.
* Patients with a history of non-adherence, who will be at risk of being unable to respect the study follow-up timetable
* Patients participating in another clinical trial within 30 days prior to inclusion
* Hb < 10 g/dL (female) or < 11g/dL (male)
* Platelets < 50 000/mm3
* Neutrophil count < 750/mm3
* Renal failure defined as creatinin clearance (MDRD) < 60ml/min
* Other antiretroviral drugs than those allowed in the study
* Contra-indications to Sofosbuvir, Ledipasvir
* Contra-indicated treatment likely to interfere with the study drugs as listed in the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2014-08; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Sustained virologic response 12 weeks after discontinuation of therapy (SVR12), i.e. at week 36. | 12 weeks post-treatment

SECONDARY OUTCOMES:
Adverse clinical and biological events that occur during the treatment and up to 24 weeks after the end of the treatment | up to 24 weeks after the end of the treatment
Number and causes of poor adherence and treatment interruptions | at 1,2,3,4,8,12,16, 20, 24 weeks during treatment, 4, 8,14,18,24 weeks after treatment discontinuationeeks after discontinuation of drugs
SVR rate 24 weeks (i.e. W48) after the end of treatment and according to the HCV sub-type | Week 48
Number of patients with HCV resistance mutations to Sofosbuvir and/or Ledipasvir | from Day(D)0 to Week (W)24
HCV viral load | at Day 0, Week 1, 2, 4, 8, 12, 16, 20, week 24, and 4, 8, 12, 18 and 24 weeks after the end of the treatment
Plasma HIV RNA levels | at Day 0, Week 4, 8, 12, 16, 20, 24, 36 and Week 48
Assess drug-drug interactions between HCV et HIV drugs | Day 0 and Week 4
  Describe pharmacokinetic parameters of HIV drugs at Day 0 and Week 4 Describe pharmacokinetic parameters of Sofosbuvir and Ledipasvir at Week 4
Patient's reported outcomes evaluation | Day 0, Week 12, Week 24 and Week 36

CONTACTS AND LOCATIONS:
Overall Officials: Eric Rosenthal, Principal Investigator — Hôpital de Nice; Eric Bellissant, Study Chair — Centre de Méthodologie et de Gestion, CHU de Rennes
Locations (1):
- Centre de Méthodologie et de Gestion de Rennes, Rennes, France